CLINICAL TRIAL: NCT02838576
Title: Effects of Hormone Replacement Therapy on Arthralgia in Postmenopausal Women: a Randomized, Double-blind Controlled Trial
Brief Title: Effects of Hormone Replacement Therapy on Arthralgia in Postmenopausal Women
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-0235
Record Dates: First submitted 2016-06-09; First posted 2016-07-20 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2019-01

CONDITIONS: Arthralgia
MeSH Terms: conditions — Arthralgia | interventions — Estrogens, Conjugated (USP); Bulk Drugs

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conjugated Equine Estrogen (Experimental): Thirty-six healthy postmenopausal women aged between 45 and 55 years will receive 0,625 mg/day conjugated equine estrogen (CEE) for 12 weeks. These 1 active pill containing conjugated equine estrogen, 0,625 mg will be provided by a laboratory with no trademark identification.
  The bottles will be numbered in code by a pharmaceutist not involved directly in study and they will donated to volunteers.
  During the intervening period, use of conjugated equine estrogen, there will be blinding. After this phase, blinding will be interrupted in order to identify volunteers who used the active drug.
  Interventions: Drug: Conjugated Equine Estrogen
- Placebo (Placebo Comparator): Thirty-six healthy postmenopausal women aged between 45 and 55 years will receive placebo pills, identical in size, shape and color to the active drug, via oral administration, for 12 weeks.
  The bottles, without trademark identification, will be numbered in code by a pharmaceutist not involved directly in study and they will donated to volunteers.
  During the intervening period, use of placebo, there will be blinding. After this phase, blinding will be interrupted in order to identify volunteers who used the active drug and placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Conjugated Equine Estrogen — Use of conjugated equine estrogen for 12 weeks. Adherence will be monitored during periodical hospital visits in order to receive pills.
  Other Names: Drug active
  Arms: Conjugated Equine Estrogen
Drug: Placebo — Use of placebo for 12 weeks. Adherence will be monitored during periodical hospital visits in order to receive pills.
  Arms: Placebo

SUMMARY:
Arthralgia has been a common complaint in postmenopausal period which seems to be involved with estrogen depletion, although, its pathophysiology isn´t completely clarified. It seems to relate with the level of physical activity, climacteric symptoms and pain catastrophizing. In view of the multiple dimensions involved in arthralgia in postmenopausal women which characterize it as a complex phenomenon, this study aims to describe the effects of hormone replacement therapy in women aged between 45 and 55 years, considering estrogen as a possible anti-nociceptive factor.

DETAILED DESCRIPTION:
This study is a randomized double-blind controlled clinical trial with postmenopausal women aged between 45 and 55 years with chronic arthralgia related to climacteric. They will be evaluated climacteric symptoms, pain intensity, level of physical activity, pain catastrophising, depression, anxiety, quality of sleep and quality of life. The volunteers will be randomized, in the proportion 1:1, to treatment with either 0,625 mg conjugated equine estrogen, via oral administration, for 12 weeks or placebo, via oral administration, for 12 weeks. The randomization will be performed by a computer-generated random numbers list. The investigators will be blinded until completion of 12 weeks. Evaluation of climacteric symptoms, pain intensity, level of physical activity, pain catastrophising, depression, anxiety, quality of sleep and quality of life will be performed in the hospital at baseline, 1, 2, 3, 6 months and 15 days. In each visit, participants will be evaluated about adverse effects such as diarrhea, nausea and vomit.

ELIGIBILITY:
Inclusion Criteria:

* age between 45 and 55 years
* chronic arthralgia related to climacteric
* regular mammography and pap smear test in the last twelve months
* availability to attend hormone replacement therapy
* maximum of ten years of amenorrhea according to the criteria of Stages of Reproductive Aging Workshop (STRAW)
* without use of hormone replacement therapy, at least, previous six months
* no contraindication to hormone replacement therapy (current or past of breast and / or cervical cancer, severe current or recent heart disease, thromboembolism, hypertension with no control, metabolic diseases (but stable thyroid disease) and endometrial hyperplasia to be enlightened
* Informed consent

Exclusion Criteria:

* autoimmune diseases
* visceral pain (chronic pelvic pain, dyspareunia, irritable bowel syndrome)
* systemic diseases (rheumatic, neurological, oncology, sexually transmitted infection)
* body mass index of 30 or greater
* soy diet
* abuse of alcohol and drugs
* large surgeries

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12-02 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Arthralgia | 6 months
  Arthralgia´ll be measured by numeric scale (0-10).

SECONDARY OUTCOMES:
Climacteric symptoms | 6 months
  Climacteric symptoms´ll be evaluated by Menopause Rating Scale - Brazilian Version. The score increases point by point with increasing severity of subjectively perceived symptoms in each of the 11 items.
Level of physical activity | 6 months
  Level of physical activity´ll be evaluated by International Physical Activity Questionnaire - Brazilian Version whose three levels of physical activity are low, moderate and high.
Pain Catastrophizing | 6 months
  Pain Catastrophizing´ll be evaluated by Pain Catastrophizing - Brazilian Version into three subscales being magnification, rumination, and helplessness. The higher the score, the more catastrophizing thoughts are present.
Health-related quality of life | 6 months
  Quality of life´ll be evaluated by Women´s Health Questionnaire - Brazilian Version (somatic symptoms, depressed mood, cognitive difficulties, anxiety and fear, sexual functioning, vasomotor symptoms, sleep problems, menstrual problems, and self-perceived attraction). The higher the score, the more pronounced the suffering and dysfunction.
Depression | 6 months
  Depression´ll be evaluated by Beck Depression Inventory - Brazilian Version. The standard cut-off scores are minimal, mild, moderate and severe depression.
Anxiety | 6 months
  Anxiety´ll be evaluated by Beck Anxiety Inventory - Brazilian Version. The standard cut-off scores are minimal, mild, moderate and severe depression.
Quality of sleep | 6 months
  Quality of sleep´ll be evaluated by Pittsburgh Sleep Quality Index - Brazilian Version. Lower scores denote a healthier sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Celeste Osório Wender, Ph.D, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Comitê de Ética em Pesquisa do Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided